CLINICAL TRIAL: NCT00400023
Title: A Phase 1, Open-Label, Randomized, Cross-Over, Pharmacokinetic Study Evaluating the Effect of the Dihydropyrimidine Dehydrogenase (Dpd) Inhibitory Action of 5-Chloro-2,4-Dihydroxypyridine (Cdhp) as an S-1 Component
Brief Title: A Phase 1, Open-Label, Randomized, Cross-Over, Pharmacokinetic Study Evaluating the Effect of S-1 on Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Peter Urrea/Senior VP Clinical and Regulatory Affairs, Taiho Pharma USA, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TPU-S1108
Record Dates: First submitted 2006-11-14; First posted 2006-11-16 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Tumors
Keywords: Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — S 1 (combination)

ARMS (2):
- 1 (Experimental): During the Cross-Over Pharmacokinetic Phase, patients will be randomly assigned to receive one of the following treatment sequences:
  * Sequence A: Single dose of 50 mg S-1 (2 capsules of 25 mg) on Day 1 followed by a single dose of 800 mg FT (8 capsules of 100 mg) on Day 8
  * Sequence B: Single dose of 800 mg FT on Day 1 followed by a single dose of 50 mg S-1 on Day 8
  Interventions: Drug: S-1
- 2 (Active Comparator): During the Cross-Over Pharmacokinetic Phase, patients will be randomly assigned to receive one of the following treatment sequences:
  * Sequence A: Single dose of 50 mg S-1 (2 capsules of 25 mg) on Day 1 followed by a single dose of 800 mg FT (8 capsules of 100 mg) on Day 8
  * Sequence B: Single dose of 800 mg FT on Day 1 followed by a single dose of 50 mg S-1 on Day 8
  Interventions: Drug: FT

INTERVENTIONS:
Drug: S-1 — During the Cross-Over PK Phase, S-1 will be administered as a 50 mg oral fixed dose and FT will be administered as an 800 mg oral fixed dose.
  During the S-1 Extension Phase (Part 2), S-1 30 mg/m2 will be administered orally BID for 2 weeks (Day 1 through Day 14) followed by a 1-week recovery period (Day 15 through Day 21). This cycle will be repeated every 3 weeks.
  Arms: 1
Drug: FT — During the Cross-Over PK Phase, S-1 will be administered as a 50 mg oral fixed dose and FT will be administered as an 800 mg oral fixed dose.
  Arms: 2

SUMMARY:
This is a Phase 1, open-label, randomized, 2-sequence, cross-over, pharmacokinetic (PK) study evaluating the effect of the DPD inhibitory action of CDHP as an S-1 component compared with FT alone on the PK of 5-FU in patients with advanced solid tumors. The study will be conducted in 2 parts (Cross-Over Pharmacokinetic Phase and S-1 Extension Phase).

ELIGIBILITY:
Inclusion Criteria:

A patient must meet all of the following inclusion criteria to be eligible for enrollment in this study:

1. Has histologically or cytologically proven advanced solid tumors for which no standard therapy exists.
2. Has provided written informed consent.
3. Is 18 years of age or older.
4. Is able to take medications orally.
5. Has Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2 (Appendix A, Performance Status).
6. Has adequate organ function as defined by the following criteria:

   * Has transaminases AST (SGOT) and ALT (SGPT) ≤ 2.5 times the upper limit of normal (ULN). If liver function abnormalities are due to underlying malignancy, then AST (SGOT) and ALT (SGPT) may be ≤ 5 times ULN.
   * Has a total serum bilirubin ≤ 1.5 times ULN.
   * Has an absolute granulocyte count ≥ 1,500/mm3 (ie, ≥ 1.5 x 109/L by International Units [IU]).
   * Has a platelet count ≥ 100,000/mm3 (IU: ≥ 100 x 109/L).
   * Has a hemoglobin value of ≥ 9.0 g/dL.
   * Has a calculated creatinine clearance > 60 mL/min (by Cockcroft-Gault formula.76 See Appendix E).
7. Is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

Exclude a patient from this study if he/she does not fulfill the inclusion criteria, or if any of the following conditions are observed:

1. Has had treatment with any of the following within the specified time frame prior to study drug administration:

   * An investigational agent received either concurrently or within the last 30 days.
   * Previous therapy for malignancy within 21 days, including any chemotherapy, immunotherapy, biologic or hormonal therapy (6 weeks for nitrosureas or mitomycin C).
   * Previous radiotherapy within 14 days.
   * Current enrollment in another clinical study with an investigational agent. Patients participating in surveys or observational studies are eligible to participate in this study.
2. Has a serious illness or medical condition(s) including, but not limited to, the following:

   * Myocardial infarction within the last 6 months, severe/unstable angina, congestive heart failure (New York Heart Association [NYHA] Class III or IV, see Appendix F).
   * Known (at the time of entry) gastrointestinal disorder, including malabsorption,chronic nausea, vomiting, or diarrhea present to the extent that it might interfere with oral intake and absorption of the study medication.
   * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study.
   * Known brain metastasis.
   * Known leptomeningeal metastasis.
   * Manifest ascites.
   * Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
3. Is receiving a concomitant treatment with drugs interacting with S-1 or FT. The following drugs are prohibited because there may be an interaction with S-1 or FT:

   * Sorivudine, uracil, dipyridamole, cimetidine and folinic acid (may enhance S-1 or FT activity).
   * Allopurinol (may diminish S-1 or FT activity).
   * Phenytoin (S-1 or FT may enhance phenytoin activity).
   * Flucytosine, a fluorinated pyrimidine antifungal agent (may enhance S-1 or FT, and flucytosine activity).
   * Pilocarpine (may inhibit CYP2A6 activity).
4. Has sensitivity to 5-FU.
5. Is a pregnant or lactating female.
6. Is a patient with reproductive potential who refuses to use an adequate means of contraception (including male patients). 3.3.3 Discontinuation Criteria Clearly document the reason for the patient's discontinuation in the patient's source documents and on the CRF. Discontinue the patient from study if any of the following occur:

   * Patient withdraws consent.
   * Patient has toxicities that, in the opinion of the Investigator, require the patient's discontinuation.
   * Patient has an intercurrent illness that in the opinion of the Investigator requires the patient's discontinuation.
   * The Investigator concludes that it is in the patient's best interest to discontinue therapy.
   * Patient is willingly or inadvertently noncompliant in the opinion of the Investigator and requires the patient to be discontinued.
   * During optional Extension Phase, the patient has objective PD (defined by imaging studies or clinical evaluation). g. During optional Extension Phase, the patient requires a recovery period of > 4 weeks (ie, more than 3 weeks from the scheduled start date of the next cycle; see Section 4.5.4.1.1).
   * The patient completes the Cross-Over Pharmacokinetic Phase but does not choose to enter the optional S-1 Extension Phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Cross-Over Pharmacokinetic Phase: To compare plasma concentrations, investigate the plasma and urine pharmacokinetic profiles, and to evaluate the duration of DPD inhibition after the administration of S-1 | The Cross-Over Pharmacokinetic phase (Part 1) will last 11 days
S-1 Extension Phase: Efficacy (antitumor response) | Each cycle of the S-1 Extension Phase (Part 2) will be 21 days (14 days S-1 treatment, 7 days recovery). The end of study for the Extension Phase will be 30 days after the last dose of S-1.
S-1 Extension Phase: Safety (Adverse events, lab assessments) | Each cycle of the S-1 Extension Phase (Part 2) will be 21 days (14 days S-1 treatment, 7 days recovery). The end of study for the Extension Phase will be 30 days after the last dose of S-1.
S-1 Extension Phase: Pharmacokinetic profiles of the components of S-1 and their metabolites, and duration of DPD inhibition after administration of multiple doses (end of Cycle 1) | Each cycle of the S-1 Extension Phase (Part 2) will be 21 days (14 days S-1 treatment, 7 days recovery). The end of study for the Extension Phase will be 30 days after the last dose of S-1.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Premiere Oncology, A Medical Corporation, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut